CLINICAL TRIAL: NCT02535715
Title: A Euglycemic Insulin Clamp Study in Type 1 Diabetic Patients With Oral Insulin (ORAMED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Oramed, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HSC20140476H
Record Dates: First submitted 2015-08-12; First posted 2015-08-31 (Estimated); Results first posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2017-05

CONDITIONS: Type 1 Diabetes
Keywords: Oral Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ORAMED ORMD-0801 capsules- 2x8mg 1st; 3x8mg 2nd, 1x16mg 3rd (Experimental): Two 8 mg ORAMED capsules containing insulin then 3X8mg ORAMED capsules containing insulin, second study then 1X16mg ORAMED capsules containing insulin, third study
  Interventions: Drug: ORMD-0801 capsules- 2x8mg; Drug: ORMD-0801 capsules- 3x8mg; Drug: ORMD-0801 capsules- 1x16mg
- ORAMED ORMD-0801 capsules- 3x8mg 1st, 1x16mg 2nd, 2x8mg 3rd (Experimental): Three 8mg ORAMED capsules containing insulin then 1X16mg ORAMED capsules containing insulin, second study then 2X8mg ORAMED capsules containing insulin, third study
  Interventions: Drug: ORMD-0801 capsules- 2x8mg; Drug: ORMD-0801 capsules- 3x8mg; Drug: ORMD-0801 capsules- 1x16mg
- ORAMED ORMD-0801 capsules-1x16mg 1st, 2x8mg 2nd, 3x8mg 3rd (Experimental): One 16mg ORAMED capsule containing insulin then 2X8mg ORAMED capsule containing insulin, second study then 3X8mg ORAMED capsule containing insulin, third study
  Interventions: Drug: ORMD-0801 capsules- 2x8mg; Drug: ORMD-0801 capsules- 3x8mg; Drug: ORMD-0801 capsules- 1x16mg

INTERVENTIONS:
Drug: ORMD-0801 capsules- 2x8mg — Participants who receive this intervention first, then receive either ORMD-0801- 3x8mg or 1x16mg dose after a 3 day to 4 week interval. Participants receiving this drug as the second drug intervention will then receive the third intervention after a 3 day to 4 week interval. ORMD-0801 capsules are an oral insulin that has shown promise in preliminary studies. Investigators will evaluate this novel insulin preparation as a potential therapeutic option in diabetic patients.
  Other Names: Oral Insulin Capsules
Drug: ORMD-0801 capsules- 3x8mg — Participants who receive this intervention first, then receive either ORMD-0801- 2x8mg or 1x16mg dose after a 3 day to 4 week interval. Participants receiving this drug as the second drug intervention will then receive the third intervention after a 3 day to 4 week interval. ORMD-0801 capsules are an oral insulin that has shown promise in preliminary studies. Investigators will evaluate this novel insulin preparation as a potential therapeutic option in diabetic patients.
  Other Names: Oral Insulin Capsules
Drug: ORMD-0801 capsules- 1x16mg — Participants who receive this intervention first, then receive either ORMD-0801- 2x8mg or 3x8mg dose after a 3 day to 4 week interval. Participants receiving this drug as the second drug intervention will then receive the third intervention after a 3 day to 4 week interval. ORMD-0801 capsules are an oral insulin that has shown promise in preliminary studies. Investigators will evaluate this novel insulin preparation as a potential therapeutic option in diabetic patients.
  Other Names: Oral Insulin Capsules

SUMMARY:
ORAMED has developed an oral insulin that, in preliminary studies, has shown promise. In the present study investigators will perform a pharmacodynamic/pharmacokinetic study to evaluate this novel insulin preparation as a potential therapeutic option in diabetic patients.

DETAILED DESCRIPTION:
Insulin therapy is an absolute requirement in type 1 diabetic patients. Multiple injections present a barrier to achieving normal/near-normal glucose control in diabetic patients (1). Therefore, there has been considerable interest in developing alternative routes of insulin administration. ORAMED has developed an oral insulin that, in preliminary studies, has shown promise. In the present study investigators will perform a pharmacodynamic/pharmacokinetic study to evaluate this novel insulin preparation as a potential therapeutic option in type 1 diabetic patients.

10 type 1 diabetic subjects will be studied.

Each subject will be studied on three occasions with an interval of 3 days to 4 weeks between each study. During each study subjects will receive one intervention at a time in random order: (i) two 8 mg ORAMED capsule containing insulin; (ii) three 8 mg ORAMED capsules containing insulin; (iii) one 16 mg ORAMED capsule containing insulin. If the fasting plasma glucose is >200mg/dl on the procedure day, the procedure will be rescheduled.

Prior to each study subjects will refrain from eating (except water) after 10 at night and report to the Clinical Research Center at approximately 7 in the morning. A catheter will be placed in an antecubital vein and a prime (40 microCuries x fasting plasma glucose/100) - continuous (0.4 microCuries/min) infusion of tritiated glucose will be started and continued until the end of the study. Plasma glucose will be monitored and if necessary during the 1st hour of tracer equilibration, a small amount of IV regular insulin will be administered to obtain a fasting plasma glucose of 100-130mg/dl. After a 3-hour tracer equilibration, subjects will ingest the ORAMED capsule containing insulin and a variable infusion of 20% glucose will be started to maintain the plasma glucose concentration between 100-120 mg/dl. Plasma samples for glucose, insulin, glucagon, and free fatty acid (FFA) concentrations and tritiated glucose radioactivity will be obtained every 5-15 minutes for 4 hours following the ingestion of the ORAMED capsule containing insulin.

Calculations: Following an overnight fast, steady state conditions prevail and the basal rate of glucose appearance equals the rate of glucose disappearance and is calculated as the tritiated glucose infusion rate divided by the tritiated glucose specific activity. Under postabsorptive conditions, Basal rate of glucose appearance primarily reflects hepatic glucose production (2). Following the ingestion of oral insulin, non-steady state conditions prevail and Ra and Rd are calculated using Steele's equation (3). Endogenous (primarily reflects liver) glucose production is calculated by subtracting the exogenous glucose infusion rate from the tracer-derived rate of glucose appearance. Endogenous rate of glucose disappearance reflects glucose uptake by all tissues in the body, but primarily reflects skeletal muscle (4).

Sample Size: The present study represents a pilot study to gain information about the absorption of oral insulin and its effect on hepatic and peripheral (skeletal muscle) glucose metabolism. This information will be used to determine whether the ORAMED oral insulin preparation represents a viable option to treat diabetic subjects, to gain information about the dose response effect of ORAMED insulin on glucose metabolism, and to provide quantitative data about the effect of oral insulin on hepatic and peripheral (muscle) glucose metabolism. Therefore, the investigators conservatively have set the sample size at 10.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18 and 70 years of age
* Must have type 1 diabetes
* Must be in good general health by routine history and physical exam
* A1c <10.0%
* BMI = 18-40 kg/m2
* On no medications known to affect glucose metabolism other than insulin
* Hematocrit ≥ 34 vol%
* Liver Function Tests < 3 x Upper Normal Limit
* Plasma creatinine < 1.8 mg/dl

Exclusion Criteria:

* Under 18 years of age and over 70 years of age
* Does not have type 1 diabetes
* A1c > 10.0%
* BMI < 18 or > 40 kg.m2
* On medications known to affect glucose metabolism other than insulin
* Hematocrit ≤ 34 vol%
* Liver Function Tests >3 x Upper Normal Limit
* Plasma creatinine > 1.8 mg/dl

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-01; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph A DeFronzo, MD, Principal Investigator — University of Texas
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Background] Polonsky WH, Fisher L, Guzman S, Villa-Caballero L, Edelman SV. Psychological insulin resistance in patients with type 2 diabetes: the scope of the problem. Diabetes Care. 2005 Oct;28(10):2543-5. doi: 10.2337/diacare.28.10.2543. No abstract available. PMID 16186296
- [Background] DeFronzo RA, Ferrannini E, Simonson DC. Fasting hyperglycemia in non-insulin-dependent diabetes mellitus: contributions of excessive hepatic glucose production and impaired tissue glucose uptake. Metabolism. 1989 Apr;38(4):387-95. doi: 10.1016/0026-0495(89)90129-7. PMID 2657323
- [Background] STEELE R. Influences of glucose loading and of injected insulin on hepatic glucose output. Ann N Y Acad Sci. 1959 Sep 25;82:420-30. doi: 10.1111/j.1749-6632.1959.tb44923.x. No abstract available. PMID 13833973

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects will be assigned to all 3 interventions during the study. One intervention will be assigned at a time, but in random order, with a 3 day to 4 week interval between interventions.
Groups:
- 2 x 8mg Oral Insulin Capsules: Subject enrolled in study who will be assigned to different interventions for the 3 periods of the study with a 3 day to 4 week interval between the different interventions. For this arm, participants will receive the 2x8mg dose first.
  2 x 8mg Oral Insulin Capsules 3 x 8mg Oral Insulin Capsules
  1 x 16mg Oral Insulin Capsule
- 3 x 8mg Oral Insulin Capsules: Subject enrolled in study who will be assigned to different interventions for the 3 periods of the study with a 3 day to 4 week interval between the different interventions. For this arm, participants will receive the 3x8mg dose first.
  2 x 8mg Oral Insulin Capsules 3 x 8mg Oral Insulin Capsules
  1 x 16mg Oral Insulin Capsule
- 1 X 16mg Oral Insulin Capsule: Subject enrolled in study who will be assigned to different interventions for the 3 periods of the study with a 3 day to 4 week interval between the different interventions. For this arm, participants will receive the 1 x 16mg dose first.
  2 x 8mg Oral Insulin Capsules 3 x 8mg Oral Insulin Capsules
  1 x 16mg Oral Insulin Capsule
Period: Overall Study
Arm/Group | 2 x 8mg Oral Insulin Capsules | 3 x 8mg Oral Insulin Capsules | 1 X 16mg Oral Insulin Capsule
Started | 4 | 4 | 3
Completed | 4 | 4 | 2
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Type 1 Diabetes Mellitus subjects in good general health
Groups:
- Overall Study: Two 8 mg ORAMED capsules containing insulin then Three 8mg ORAMED capsules containing insulin then One 16mg ORAMED capsules containing insulin
  ORMD-0801 capsules: ORMD-0801 capsules are an oral insulin that has shown promise in preliminary studies. Investigators will evaluate this novel insulin preparation as a potential therapeutic option in diabetic patients.
Arm/Group | Overall Study
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian or Pacific Islander | 1
  Black-non Hispanic | 1
  Hispanic | 3
  White non-Hispanic | 6
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Hepatic Glucose Production (Co-primary Outcome)
Description: Tritiated glucose infusion during procedures (Baseline and every 30 minutes during procedures) Calculated from plasma(mg/kg-minute). Averaged every 30 minutes.
Time Frame: Participants will be followed during the procedures, until all 3 procedures are completed, an average of 1 month
Measure: Mean (Standard Error); unit: mg/kg-minute
Groups:
- 2X 8mg Oral Insulin Capsules: ORAMED provided 8 mg oral insulin capsules. Two (2) capsules administered at time 0 of the euglycemic clamp
- 3X 8mg Oral Insulin Capsules: ORAMED provided 8 mg oral insulin capsules. Three (3) capsules administered at time 0 of the euglycemic clamp
- 1X 16mg Oral Insulin Capsules: ORAMED provided 16mg oral insulin capsules. One(1) capsule administered at time 0 of the euglycemic clamp
Arm/Group | 2X 8mg Oral Insulin Capsules | 3X 8mg Oral Insulin Capsules | 1X 16mg Oral Insulin Capsules
Number analyzed (Participants) | 11 | 11 | 10
mg/kg-minute
  -180 to 0 | 2.0 (0.1) | 2.0 (0.1) | 2.1 (0.3)
  1-30 minutes | 1.8 (0.2) | 1.9 (0.1) | 2.1 (0.3)
  31-60 minutes | 1.6 (0.2) | 1.7 (0.20) | 2.1 (0.4)
  61-90 minutes | 1.5 (0.2) | 1.6 (0.1) | 1.9 (0.4)
  91-120 minutes | 1.6 (0.2) | 1.7 (0.2) | 1.7 (0.5)
  121-150 minutes | 1.5 (0.2) | 1.6 (0.2) | 1.6 (0.5)
  151-180 minutes | 1.6 (0.2) | 1.6 (0.2) | 1.7 (0.5)
  181-210 minutes | 1.5 (0.2) | 1.5 (0.2) | 1.4 (0.2)
  211-240 | 1.4 (0.2) | 1.5 (0.2) | 1.5 (0.3)

2. Secondary Outcome: Plasma Insulin Concentrations
Description: Baseline and every 15 minutes during procedures (microIU/mL).
Time Frame: Participants will be followed during the procedures, until all 3 procedures are completed, an average of 1 month
Population: Plasma insulin Concentrations were measured during each procedure in a type 1 DM population Analysis from one subject was not included: Results below threshold of assay
Measure: Mean (Standard Deviation); unit: microUnits/mL
Groups:
- Two 8mg ORAMED Capsules Containing Insulin: Two (2) 8 mg ORAMED capsules containing insulin
  ORMD-0801 capsules: ORMD-0801 capsules are an oral insulin that has shown promise in preliminary studies. Investigators will evaluate this novel insulin preparation as a potential therapeutic option in diabetic patients.
- Three 8mg ORAMED Capsules: Three (3) 8mg ORAMED INSULIN CAPSULES containing oral insulin
- One 16mg ORAMED Capsule: One (1) 16mg ORAMED INSULIN CAPSULE containing oral insulin
Arm/Group | Two 8mg ORAMED Capsules Containing Insulin | Three 8mg ORAMED Capsules | One 16mg ORAMED Capsule
Number analyzed (Participants) | 11 | 11 | 10
microUnits/mL
  Baseline | 9 (4) | 8 (8) | 7 (4)
  15 minutes | 9 (4) | 8 (6) | 7 (6)
  30 minutes | 8 (5) | 8 (6) | 8 (6)
  45 minutes | 8 (4) | 7 (6) | 7 (5)
  60 minutes | 8 (5) | 8 (6) | 7 (4)
  75 minutes | 8 (5) | 8 (6) | 7 (5)
  90 minutes | 9 (4) | 8 (6) | 7 (5)
  105 minutes | 9 (6) | 8 (6) | 7 (5)
  120 minutes | 9 (6) | 8 (5) | 7 (6)
  135 minutes | 8 (5) | 8 (5) | 7 (6)
  150 minutes | 8 (5) | 8 (5) | 7 (5)
  165 minutes | 9 (6) | 8 (5) | 6 (4)
  180 minutes | 9 (6) | 8 (6) | 6 (4)
  195 minutes | 9 (6) | 8 (6) | 6 (4)
  210 minutes | 8 (5) | 8 (6) | 6 (5)
  230 minutes | 9 (6) | 8 (6) | 7 (4)
  240 minutes | 9 (6) | 7 (6) | 7 (4)

3. Secondary Outcome: Plasma Glucose Concentrations
Description: Measured at baseline and every 5 minutes during the procedures(mg/dL), Averaged over 30 minute intervals during the procedure
Time Frame: Participants will be followed during the procedures, until all 3 procedures are completed, an average of 1 month
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Two 8mg ORAMED Capsules Containing Insulin | Three 8mg ORAMED Capsules | One 16mg ORAMED Capsule
Number analyzed (Participants) | 10 | 10 | 10
mg/dl
  -180 to 0 | 109 (9) | 120 (10) | 123 (8)
  1-30 minutes | 98 (5) | 110 (8) | 115 (7)
  31-60 minutes | 98 (5) | 113 (7) | 116 (6)
  61-90 minutes | 100 (6) | 118 (8) | 116 (5)
  91-120 minutes | 103 (5) | 117 (9) | 115 (5)
  121 to 150 minutes | 105 (5) | 115 (8) | 118 (6)
  151 to 180 minutes | 107 (5) | 113 (8) | 120 (7)
  181 to 210 minutes | 110 (6) | 112 (9) | 122 (8)
  210 to 240 minutes | 111 (7) | 117 (10) | 128 (8)

4. Secondary Outcome: Plasma Glucagon Concentrations
Description: Measured at baseline and every 30 minutes during the procedures (pg/mL)
Time Frame: Participants will be followed during the procedures, until all 3 procedures are completed, an average of 1 month
Population: Glucagon measured by RIA kit, EMD Millipore.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | 2X 8mg Oral Insulin Capsules | 3X 8mg Oral Insulin Capsules | 1X 16mg Oral Insulin Capsules
Number analyzed (Participants) | 11 | 11 | 10
pg/mL
  -180 to 0 minutes | 29 (4) | 37 (4) | 37 (4)
  1-30 minutes | 29 (4) | 38 (5) | 36 (4)
  31-60 minutes | 27 (3) | 37 (4) | 34 (5)
  61-90 minutes | 29 (3) | 36 (4) | 34 (5)
  91-120 minutes | 28 (4) | 34 (4) | 33 (4)
  121-150 minutes | 26 (3) | 35 (4) | 34 (4)
  151-180 minutes | 26 (4) | 35 (4) | 33 (4)
  181 to 210 minutes | 23 (3) | 35 (4) | 31 (4)
  211-240 minutes | 24 (3) | 36 (4) | 32 (4)

5. Secondary Outcome: Plasma Free Fatty Acid Concentrations
Description: Measured at baseline and every 30 minutes during the procedures (micro mol/L)
Time Frame: Participants will be followed during the procedures, until all 3 procedures are completed, an average of 1 month
Population: Wako Calorometric
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | 2X 8mg Oral Insulin Capsules | 3X 8mg Oral Insulin Capsules | 1X 16mg Oral Insulin Capsules
Number analyzed (Participants) | 10 | 10 | 10
mmol/L
  Baseline | 380 (68) | 402 (80) | 410 (87)
  1-30 minutes | 408 (76) | 465 (81) | 467 (69)
  31-60 minutes | 463 (78) | 533 (96) | 448 (61)
  61-90 minutes | 472 (74) | 545 (102) | 489 (63)
  91-120 minutes | 495 (84) | 473 (94) | 506 (56)
  121-150 minutes | 528 (74) | 501 (97) | 509 (54)
  151-180 minutes | 547 (80) | 486 (95) | 545 (53)
  181-210 minutes | 523 (75) | 485 (97) | 533 (63)
  211-240 minutes | 490 (69) | 486 (95) | 538 (74)
Statistical Analysis 1: Comparison: 2X 8mg Oral Insulin Capsules vs 3X 8mg Oral Insulin Capsules vs 1X 16mg Oral Insulin Capsules; Test type: Superiority — ANOVA Bonferroni adjustment; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over period of participation of each subject: From signing of informed consent, including between procedures, until conclusion of 3rd procedure. Subjects were instructed to call us if any adverse events after this timeframe.
Groups:
- 2X 8mg Capsules: Adverse event reporting for subjects during the 2X 8mg dosing regimen
- 3X 8mg Oral Insulin Capsules: Adverse event reporting for subjects during the 3X 8mg dosing regimen
- 1X 16mg Capsules: Adverse event reporting for subjects during the 1X 16mg dosing regimen
Arm/Group | 2X 8mg Capsules | 3X 8mg Oral Insulin Capsules | 1X 16mg Capsules
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 1/11 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2X 8mg Capsules (N=11) | 3X 8mg Oral Insulin Capsules (N=11) | 1X 16mg Capsules (N=10)
Hypoglycemia (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT02535715/Prot_SAP_000.pdf